CLINICAL TRIAL: NCT03107312
Title: Bioarray Compilation for the Serological Assessment of Immunity Against Vaccine-preventable Infections of Available Prophylaxis in Refugees and Immigrants
Brief Title: Bioarray for the Serological Assessment of Immunity Against Vaccine-preventable Infections
Acronym: StikoSero
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Jena University Hospital (Other)
Responsible Party: Principal Investigator, Mathias Pletz, Director, Center for Infectious Diseass and Infection Control, Jena University Hospital
Other Study IDs: StikoSero
Record Dates: First submitted 2017-04-05; First posted 2017-04-11 (Actual); Last update posted 2017-05-15 (Actual); Status verified 2017-05

CONDITIONS: Immunization; Infection
MeSH Terms: conditions — Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Known vaccination history: Single blood sample collection from subjects with verified records of vaccination or recent booster immunization against measles, mumps, rubella, varicella, tetanus, pertussis, poliomyelitis, diphtheria, meningococcal infection
  Interventions: Procedure: Single blood sample collection
- Migrants: Single blood sample collection from recent migrants to Germany without verified vaccination records
  Interventions: Procedure: Single blood sample collection

INTERVENTIONS:
Procedure: Single blood sample collection — Collection of single blood sample of 10 ml volume by venepuncture

SUMMARY:
Recent observations in Germany revealed above-average high proportions of refugees affected by infectious diseases of public health significance. Scrutiny of the vaccination status showed sizeable presence of seronegative subjects, with conspicuously higher prevalence among children and adolescents, thus indicating urgent necessity of i) rapid identification of carriers of vaccine-preventable diseases and ii) adjustment of protection against such infections to European Standards. Rapid immune status check needs comprehensive diagnostic tool permitting simultaneous assessment of seropositivity. Validation of such tools requires comparisons of the immune status of subjects with known vaccination history with that of migrants with incomplete or missing health and vaccination records.

DETAILED DESCRIPTION:
The current massive inflow of refugees and migrants poses urgent necessity of i) rapid identification of carriers of communicable diseases and ii) adjustment of protection against vaccine-preventable infections to European standards. While universal vaccination is supposed to ensure the intended degree of protection, targeted vaccination on the basis of previous assessment of the immune status (seropositivity) was repeatedly shown to be a cost-efficient alternative. Currently, the broad use of immune status assessment prior to targeted vaccination is impeded by the necessity to apply separate seropositivity detection assays for each individual condition. This drawback can be overcome by the introduction of a comprehensive diagnostic tool permitting simultaneous assessment of seropositivity for several vaccine-preventable infections.

The objective of the present study consists in compilation of an array of sera from

* subjects with known history of immunization against vaccine-preventable infections for which vaccines are routinely available (measles, mumps, rubella, varicella, tetanus, pertussis, poliomyelitis, diphtheria, meningococcal infection) and
* new migrants/refugees without reliable vaccination records and undefined immune status to be subsequently used for the validation of a multi-pronged diagnostic tool for seropositivity detection

ELIGIBILITY:
Inclusion Criteria:

* Age above 18 years
* Signed informed consent

Exclusion Criteria:

* Acute infectious condition
* Glucocorticoid medication above 0.3 mg/kg Prednisolone equivalent over the preceding 30 days
* Treatment with recognized T cell immunosuppressant or nucleoside analogues during the preceding 90 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects with verified/complete or non-verified/incomplete vaccination history
Sampling Method: Non-Probability Sample
Enrollment: 900 (Estimated)
Dates: Start 2017-04-01 (Actual); Primary Completion 2018-03-31 (Estimated); Study Completion 2018-03-31 (Estimated)

PRIMARY OUTCOMES:
Serum sample array compilation | 1 year
  Collection of individual serum samples from participants with different vaccination history

CONTACTS AND LOCATIONS:
Overall Officials: Mathias Pletz, M.D., Principal Investigator — Center for Infectious Diseases and Infection Control
Locations (1):
- Center for Infectious Diseases and Infection Control, Jena University Hospital, Jena, Thuringia, Germany

IPD SHARING:
Plan to Share IPD: No